CLINICAL TRIAL: NCT05807620
Title: A Clinical Study to Evaluate the Efficacy and Tolerability of an Eye Cream for Moderate to Severe Dark Circles and Undereye Puffiness
Brief Title: A 12 Week Study to Evaluate the Efficacy of an Eye Cream
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Revision Skincare (Industry)
Collaborators: Validated Claim Support (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS211024
Record Dates: First submitted 2023-03-20; First posted 2023-04-11 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Periorbital Hyperpigmentation; Periorbital Edema; Fine Lines; Wrinkle
Keywords: dark circles; puffiness; brightening
MeSH Terms: conditions — Orbital Cellulitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eye Cream (Experimental): Eye Cream composed of botanical extracts, bioavailable peptides, THD Ascorbate and Caffeine.
  Subjects to apply a dime size amount onto the under-eye area and crow's feet area while avoiding direct eye contact twice daily for the duration of the 12-week clinical study.
  Interventions: Other: Gentle Cleansing Lotion; Other: Facial Moisturizer; Other: Sunscreen SPF 30

INTERVENTIONS:
Other: Gentle Cleansing Lotion — Facial cleansing lotion to be used by study participants (morning and evening, 2x daily).
Other: Facial Moisturizer — Anti-aging facial moisturizer to be used by study participants after anti-aging daily serum before sunscreen (morning and evening, 2x daily).
Other: Sunscreen SPF 30 — Neutrogena Ultra Sheer Dry Touch SPF 30. Sunscreen to be applied after application of the facial moisturizer in the morning. Participants were asked to reapply every 2 hours.
  Per FDA this intervention is an over the counter

SUMMARY:
This single center, open-label clinical study was conducted to assess the efficacy and tolerance of a topical eye cream when used over the course of 12 weeks by healthy women with moderate to severe under-eye dark circles, moderate under eye puffiness, and mild fine lines and wrinkles. A total of 37 subjects were enrolled into the study.

DETAILED DESCRIPTION:
This single center, open-label clinical study was conducted to evaluate the efficacy and tolerability of an eye cream on healthy female subjects between 35 to 60 years of age with Fitzpatrick Skin Type I - VI, and moderate to severe dark circles and under-eye puffiness. This study aims to evaluate the following objectives:

1. To evaluate the eye cream impact on undereye dark circles, undereye puffiness, fine lines and wrinkles periorbital eye area, and overall appearance periorbital eye area, as evaluated by investigator clinical grading, chromameter, VISIA clinical photography, and subjective questionnaire performed at baseline, week 4, week 8, and week 12.
2. To evaluate the eye cream impact on under eye blood flow, as evaluated by laser doppler performed at baseline, week 8, and week 12.
3. To assess objective and subjective tolerability of Dryness, Erythema, and Edema, and Burning, Stinging, Peeling, and Itching evaluated by investigator and subjective grading at baseline, week 4, week 8, and week 12.

A total of 37 subjects completed the study.

ELIGIBILITY:
Inclusion Criteria:

* Females in good general health
* With Fitzpatrick Skin Type I - VI
* Moderate to severe under eye dark circles
* Moderate undereye puffiness
* Mild to moderate fine lines and wrinkles

Exclusion Criteria:

* Subjects who have used retinol or eye cream / serum 7 days prior to study commencement
* Nursing, pregnant, or planning a pregnancy during this study
* Having a health condition and / or pre-existing or dormant dermatologic disease on the face

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Change in Investigator Clinical Grading versus Baseline | 12 weeks
  The primary efficacy endpoint will be investigator clinical grading using a Modified Griffiths 10 point scale and a validated photonumeric scale for undereye dark circles
  A decrease in scores at post baseline timepoints (weeks 4, 8, and 12) in comparison to baseline indicates an improvement for the indicated parameter.
  The efficacy parameters will be assessed globally on each subject's face using a validated photonumeric scale for dark circles and Modified Griffiths 10-point scale according to the following numerical definitions (half-point scores may be used as necessary to more accurately describe the skin condition):
  0 = none (best possible condition); 1 to 3 = mild; 4 to 6 = moderate; 7 to 9 = severe (worst possible condition). The lower the score equates to the best possible outcome.
Bioinstrumentation: Laser Doppler | 12 weeks
  Bioinstrumentation measurements includes INL 191 Blood FlowMeter laser doppler
  A standard surface probe approximately 17mm in diameter was placed on the right or left undereye area per randomization and measurements in perfusion units (AU) were obtained at baseline week 8 and week 12.
  An increase in AU values indicates an improvement in dark circles
Bioinstrumentation: Chromameter | 12 weeks
  Bioinstrumentation measurements includes Chroma Meter CR-200 (Konica Minolta, Tokyo, JPN)
  Measurements were taken on the right or left undereye area, per randomization on each subject in triplicate and averaged at baseline, week 4, 8 and 12. Three color value characteristics are evaluated: L* (100 = white, 0 = black) and a* (red-green)
  An increase in L* indicates an improvement A decrease in a* indicates an improvement

SECONDARY OUTCOMES:
Lack of significant increase in objective investigator tolerability parameters at week 4, 8, and 12 compared to baseline | 12 weeks
  The second outcome measure is objective tolerability endpoint. Investigator Tolerability Assessment includes Erythema, Edema and Dryness.
  A decrease in scores or lack of significant increase at week 4, 8, and 12 in comparison to Baseline indicates tolerability/safety of the test material. Five point scale with a lower score indicating a better outcome.
  Example for Erythema: Erythema 0 = None No erythema of the treatment area
  1. = very slight erythema (barely perceptible)
  2. = well-defined erythema
  3. = Moderate to severe erythema
  4. = Severe erythema (beet redness) to slight eschar formation
Lack of significant increase in Subjective investigator tolerability parameters at week 4, 8, and 12 compared to baseline | 12 weeks
  The secondary tolerability endpoint will be the Subjective Tolerability Assessment of Stinging, Tingling, Itching, and Burning
  A decrease in scores or lack of significant increase at week 4, 8, and 12 in comparison to Baseline indicates tolerability/safety of the test material. Four point scale with a lower score indicating a better outcome.
  Example Burning.
  0 = None
  1. = Mild
  2. = Moderate
  3. = Severe

OTHER OUTCOMES:
Change In Facial parameters in a self-assessment questionnaire versus Baseline and % Agreement | 12 weeks
  Self-Assessment Questionnaire and the Subject Treatment Satisfaction. A decrease or increase in response values at week 4, 8, and 12, and indicates an improvement compared to baseline response values.
  Subjects are asked to rate based on a scoring system of the following:
  from 5 (completely agree) to 1 (completely disagree). The best outcome is to Completely Agree with the statement/ question being asked.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Hardy, Study Director — Validated Claim Support
Locations (1):
- Validated Claim Support, LLC, Teaneck, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers